CLINICAL TRIAL: NCT02936297
Title: Quantitative Measurement of Stool and Urine Gluten Immunogenic Peptides in Patients With Non-celiac Gluten Sensitivity and Healthy Patients: A Placebo-controlled Study Study
Brief Title: Gluten Ingestion Biomarkers in Patients w Gluten Sensitivity and Healthy Controls Peptides in Patients With Non-celiac Gluten Sensitivity and Healthy Patients: A Placebo-controlled Study
Acronym: NCGS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: IRB#16D.244
Record Dates: First submitted 2016-09-02; First posted 2016-10-18 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Non Celiac Gluten Sensitivity
MeSH Terms: interventions — Glutens

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lactose free placebo (Placebo Comparator): Lactose free placebo pill
  Interventions: Dietary Supplement: Lactose free placebo
- Low dose Gluten (0.5g) (Active Comparator): Low dose gluten pill
  Interventions: Dietary Supplement: Low dose Gluten
- High Dose Gluten (2.0g) (Active Comparator): High dose gluten pill
  Interventions: Dietary Supplement: High dose Gluten

INTERVENTIONS:
Dietary Supplement: High dose Gluten
  Arms: High Dose Gluten (2.0g)
Dietary Supplement: Low dose Gluten
  Arms: Low dose Gluten (0.5g)
Dietary Supplement: Lactose free placebo
  Arms: Lactose free placebo

SUMMARY:
Non-celiac gluten sensitivity (NCGS) is an emerging clinical entity defined as the presence of intestinal and/or extraintestinal symptoms induced by the ingestion or gluten and relieved by a gluten free diet (GFD) in patients without celiac disease or wheat allergy. The pathologic mechanism of the disorder is unknown, and there are no known biomarkers or associated histopathologic findings. In this prospective, randomized controlled trail, we are investigating the utility of patient reported symptom questionnaires, as well as stool gluten and urine quantification tools in patients with NCGS and healthy controls.

ELIGIBILITY:
Inclusion criteria include

* Patients > 18 years of age
* Patients willing to maintain gluten free diet for 6 weeks

Exclusion Criteria (NCGS):

* Patients < 18 years of age
* Patients with positive serology suggestive of celiac disease and/or biopsy-proven celiac disease and/or Human leukocyte antigen (HLA) DQ2 or DQ8 positivity.
* Patients with a diagnosis of inflammatory bowel disease
* Patients with a diagnosis of acute gastroenteritis
* Patients who are pregnant
* Type 1 Diabetes Mellitus

Exclusion criteria (healthy controls):

* NCGS
* Celiac disease
* Inflammatory bowel disease
* Irritable bowel syndrome
* Acute gastroenteritis
* Patients who are pregnant
* Type 1 Diabetes Mellitus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-06; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Patient estimated gluten intake after administration of gluten compared to baseline level on GFD, using the Celiac Dietary Adherence Test (CDAT) | 12 weeks
NCGS symptoms, using the Celiac Symptom Index (CSI)10 after administration of gluten compared to baseline level on GFD | 12 weeks
Stool gluten immunogenic peptides (GIP) level after administration of gluten compared to baseline level on GFD. | 12 weeks
Urine gluten immunogenic peptides (GIP) level after administration of gluten compared to baseline level on GFD | 12 weeks
Patient Estimation of Gluten Intake captured via (PEGI) questionnaire | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States